CLINICAL TRIAL: NCT05333510
Title: A Comparative Evaluation of Thromboelastography Versus Thromboelastometry for Coagulopathy Correction in Patients of Liver Cirrhosis With Non Variceal Bleed- Prospective Observational Study
Brief Title: A Comparative Evaluation of TEG Versus ROTEM for Coagulopathy Correction
Status: Completed | Type: Observational
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Other Study IDs: IEC/2021/86/MA06
Record Dates: First submitted 2022-01-13; First posted 2022-04-19 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2022-01

CONDITIONS: Liver Cirrhosis
Keywords: THROMBOELASTOGRAPHY; THROMBOELASTOMETRY; nonvariceal; bleeding
MeSH Terms: conditions — Liver Cirrhosis; Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- TEG group: Thromboelastography guided blood product administration in patients of liver cirrhosis with non variceal bleed
- ROTEM group: Throboelastometry guided blood product administration in patients of liver cirrhosis with non variceal bleed

SUMMARY:
Studies comparing Thromboelastography or Rotational thromboelastometry versus standard coagulation tests are abundant. Data comparing the two exclusively in a liver intensive care set up is limited.

Studies show that TEG and ROTEM cannot be used interchangeably in trauma, liver transplant patients, but there is limited evidence of the same in critically ill cirrhotic patients.

In this study, the investigators tried to demonstrate the comparison of blood products used to treat coagulopathy based on TEG versus ROTEM algorithms in cirrhotic patients presenting with non variceal bleeding

DETAILED DESCRIPTION:
Thromboelastography (TEG) and thromboelastometry( ROTEM) are point-of-care, global hemostasis assessment tests that measure the viscoelastic changes that occur during the hemostatic process.

Patients with cirrhosis have an imbalance of procoagulants and anticoagulants combined with alterations in fibrinolysis ,platelet number and function.

Point of care viscoelastic tests (TEG ,ROTEM) demonstrate specific functional coagulation defects that can direct blood component transfusion therapy in cirrhosis, with clinical validation of individual parameters.

Studies comparing Thromboelastography or Rotational thromboelastometry versus standard coagulation tests are abundant. Data comparing the two exclusively in a liver intensive care set up is limited.

Studies show that TEG and ROTEM cannot be used interchangeably in trauma, liver transplant patients, but there is limited evidence of the same in critically ill cirrhotic patients.

In this study, the investigators tried to demonstrate the comparison of blood products used to treat coagulopathy based on TEG versus ROTEM algorithms in cirrhotic patients presenting with non variceal bleeding

ELIGIBILITY:
Inclusion Criteria:

* patients of liver cirrhosis with non variceal bleed

Exclusion Criteria:

1. Pregnant and postpartum patients
2. died within the first 24hours of admission.
3. variceal and postvariceal ligation ulcer bleed.
4. On anticoagulants or antiplatelets at the time of admission in ICU
5. Transfusion with blood products before admission to the ICU.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients of liver cirrhosis who are presenting with non variceal bleed would be included in this study
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-01-08 (Actual); Study Completion 2022-01-08 (Actual)

PRIMARY OUTCOMES:
Total amount of blood products transfused at 8 hours(FFP, Cryoprecipitate, platelets) will be measured | 8 hours
  Total amount of blood products transfused at 8 hours(FFP, Cryoprecipitate, platelets) will be measured

SECONDARY OUTCOMES:
R time of thromboelastography | 8 hours
  R time measures time to start forming clot
K time of thromboelastography | 8 hours
  K time represents time until clot reaches a fixed strength
alpha angle of thromboelastography | 8 hours
  alpha angle represents speed of fibrin accumulation
Maximum amplitude of thromboleastography | 8 hours
  It represents the highest vertical amplitude of thromboelastography
LY30 Iin thromboelastometry | 8 hours
  It represents the percentage of amplitude reduction 30 minutes after reaching maximum amplitude
Clotting time in thromboelastometry | 8 hours
  It represents the time to start forming clot and initial fibrin formation
Clot formation time in thromboelastometry | 8 hours
  It represents the clot strengthening and rapidity of fibrin build up
Maximum clot firmness in thromboelastometry | 8 hours
  It represents the highest vertical amplitude of the thromboelastometry graph and represents clot strength
LI30 in thromboelastometry | 8 hours
  It represents clot breakdown and fibrinolysis at fixed time
Control of bleeding at 48 hours | 48 hours
  The investigators would measure the hemoglobin levels to see for any drop in concentration of hemoglobin

CONTACTS AND LOCATIONS:
Overall Officials: NIMI GOPAL, Principal Investigator — Institute of Liver and Biliary Sciences
Locations (1):
- Institute of Liver and Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Premkumar M, Saxena P, Rangegowda D, Baweja S, Mirza R, Jain P, Bhatia P, Kumar G, Bihari C, Kalal C, Vyas T, Choudhury A, Sarin SK. Coagulation failure is associated with bleeding events and clinical outcome during systemic inflammatory response and sepsis in acute-on-chronic liver failure: An observational cohort study. Liver Int. 2019 Apr;39(4):694-704. doi: 10.1111/liv.14034. Epub 2019 Feb 7. PMID 30589495
- [Background] Kumar M, Ahmad J, Maiwall R, Choudhury A, Bajpai M, Mitra LG, Saluja V, Mohan Agarwal P, Bihari C, Shasthry SM, Jindal A, Bhardwaj A, Kumar G, Sarin SK. Thromboelastography-Guided Blood Component Use in Patients With Cirrhosis With Nonvariceal Bleeding: A Randomized Controlled Trial. Hepatology. 2020 Jan;71(1):235-246. doi: 10.1002/hep.30794. Epub 2019 Aug 27. PMID 31148204
- [Background] Wikkelso A, Wetterslev J, Moller AM, Afshari A. Thromboelastography (TEG) or thromboelastometry (ROTEM) to monitor haemostatic treatment versus usual care in adults or children with bleeding. Cochrane Database Syst Rev. 2016 Aug 22;2016(8):CD007871. doi: 10.1002/14651858.CD007871.pub3. PMID 27552162
- [Background] Singh SA, Krishnan G, Ashraf H, Subramanian R, Pandey V, Nasa VK, Goyal S, Gupta S. Correlation between thromboelastography and rotational thromboelastometry values in adult liver transplant recipients. Indian J Anaesth. 2020 Apr;64(4):286-291. doi: 10.4103/ija.IJA_762_19. Epub 2020 Mar 28. PMID 32489202